CLINICAL TRIAL: NCT04376632
Title: Comparison of Health Effects of Diets With and Without Pecans
Brief Title: Diets Enriched With Pecans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Georgia Pecan Commission (Unknown)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Associate Professor, Dept. of Foods and Nutrition, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00005985
Record Dates: First submitted 2020-04-30; First posted 2020-05-06 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Hypercholesterolemia; Obesity
MeSH Terms: conditions — Hypercholesterolemia; Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are unaware that there are 2 pecan groups (with and without dietary substitution instructions)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in this group avoid all nuts for 8 weeks.
- Pecan ADD (Experimental): Participants in this group consume 68 g of pecans/d with no additional dietary instructions and avoid all other nuts.
  Interventions: Dietary Supplement: Pecan ADD
- Pecan SUB (Experimental): Participants in this group consume 68 g of pecans/d with instructions to substitute pecans with isocaloric foods in the habitual diet. They are also instructed to avoid all other nuts.
  Interventions: Dietary Supplement: Pecan SUB

INTERVENTIONS:
Dietary Supplement: Pecan ADD — Raw pecan halves without dietary substitution instructions
  Other Names: Pecan
  Arms: Pecan ADD
Dietary Supplement: Pecan SUB — Raw pecan halves with instructions to substitute pecans with isocaloric foods in the habitual diet
  Other Names: Pecan
  Arms: Pecan SUB

SUMMARY:
Background: Previous studies report that daily pecan consumption reduces cholesterol in healthy adults while promoting weight maintenance.

Purpose: To examine the impact of daily pecan consumption with and without dietary substitution instructions for an 8-week period on markers of health in adults at risk for cardiovascular disease.

DETAILED DESCRIPTION:
This was a single-blind, randomized controlled trial. The investigators recruited subjects with hypercholesterolemia (high blood cholesterol levels) or at higher risk for cardiovascular disease (CVD) (BMI > 28 kg/m2). Subjects were randomized into one of three groups: (1) the no nut group (CON), (2) pecan ADD (no diet instructions), and (3) pecan SUB (instructions to substitute pecans with isocaloric foods in habitual diet).

There was a screening visit and 3 testing visits: Baseline (visit 1), mid-visit at week 4 (visit 2), and post-visit at week 8 (visit 3). Anthropometrics, questionnaires, and a fasting blood sample were collected at each visit. A subset of participants participated in a saturated fatty acid meal challenge in which additional blood and metabolism measurements were collected.

Hypothesis: The investigators hypothesized that daily pecan consumption would result in significantly greater improvements in blood lipids, metabolism, and appetite compared to the control group. The investigators also hypothesized that pecan ADD group will result in a larger increase in body weight compared to the pecan SUB and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30-75y with higher cholesterol levels or BMI of 28 kg/m2 or greater (A higher cholesterol level is indicated by "Borderline High/Undesirable" in two or more of the variables (total cholesterol 200-239 mg/dL, LDL cholesterol 130-159 mg/dL, triglycerides 150-199 mg/dL) or "High" in either total cholesterol (240 mg/dL and higher) or LDL (160 mg/dL or higher).

Exclusion Criteria:

* Familial hypercholesterolemia (individuals with LDL levels greater than the 95th percentile or HDL levels lower than the 20th percentile based on age and sex)
* Nut consumption >2 servings/week or tree nut butter consumption >3 servings/week
* Hormone replacement therapy <5 years
* Women who are pregnant or planning to become pregnant
* Regular exercise of >3 hours/week
* Weight gain or loss of >5% of body weight during last 3 months
* Plans to begin a weight loss/exercise regiment
* History of medical or surgical events that could affect digestion or swallowing
* Gastrointestinal surgeries, conditions or disorders
* Chronic or metabolic diseases
* Atherosclerosis, previous myocardial infarction, stroke, cancer
* Fasting blood glucose levels >126 mg/dl
* Blood pressure >180/120 mmHg
* Medication use that affects digestion, absorption, metabolism
* Lipid-lowering medications
* Medications for diabetes or attention deficit disorders (with or without hyperactivity)
* Steroid/hormone therapies
* Individuals on medically prescribed or special diet
* Individuals with food allergies to foods specifically in the study
* Individuals taking fish oil supplements
* Excessive alcohol consumption (greater than 3 drinks/d for men; greater than 2 drinks/d for women)
* Tobacco or nicotine use

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Change in baseline fasting blood lipids at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Total cholesterol (mg/dL), high-density lipoprotein (HDL) cholesterol (mg/dL), triglycerides (mg/dL), low-density lipoprotein (LDL) cholesterol (mg/dL), non-HDL cholesterol (mg/dL), apolipoprotein B (mg/dL)
Change in baseline lipoprotein(a), lipoprotein particle number, and lipoprotein size at 4 and 8 weeks | Baseline, 4 weeks, 8 weeks
  Low-density lipoprotein (LDL) particle number (nmol/L), LDL small (nmol/L), LDL medium (nmol/L), HDL large (nmol/L), lipoprotein(a) (nmol/L)
Change in baseline low-density lipoprotein (LDL) peak size at 4 and 8 weeks | Baseline, 4 weeks, 8 weeks
  LDL peak size (angstrom)
Change in baseline weight at 4 and 8 weeks | Baseline, 4 weeks, 8 weeks
  Weight (kg)
Change in baseline waist and hip circumference at 4 and 8 weeks | Baseline, 4 weeks, 8 weeks
  waist and hip circumference (cm)
Change in baseline total body fat percentage at 4 and 8 weeks | Baseline, 4 weeks, 8 weeks
  Total body fat percentage (%)

SECONDARY OUTCOMES:
Change in fasting and postprandial peptide YY, cholecystokinin (CCK), and ghrelin from baseline to 8 weeks | Data will be collected at fasting at baseline, 4 weeks and 8 weeks. Postprandial data will be collected at baseline and 8 weeks.
  Peptide YY (pg/mL), CCK (pg/mL) and ghrelin (pg/mL)
Change in fasting and postprandial glucose and triglycerides from baseline to 8 weeks | Data will be collected at fasting at baseline, 4 weeks and 8 weeks. Postprandial data will be collected at baseline and 8 weeks.
  Glucose (mg/dL) and triglycerides (mg/dL)
Change in fasting and postprandial non-esterified free fatty acids (NEFA) from baseline to 8 weeks | Data will be collected at fasting at baseline, 4 weeks and 8 weeks. Postprandial data will be collected at baseline and 8 weeks.
  NEFA (mEq/L)
Change in fasting and postprandial insulin from baseline to 8 weeks | Data will be collected at fasting at baseline, 4 weeks and 8 weeks. Postprandial data will be collected at baseline and 8 weeks.
  Insulin (uU/mL)
Change in resting metabolic rate (RMR) from baseline to 8 weeks | Baseline and 8 weeks
  RMR (kcals/d) measured via indirect calorimetry
Change in diet induced thermogenesis (DIT) from baseline to 8 weeks | Baseline and 8 weeks
  DIT (kcals) measured via indirect calorimetry
Change in fasting and postprandial carbohydrate and fat oxidation from baseline to 8 weeks | Measured at fasting and for 3.5h postprandially at baseline and 8 weeks
  Carbohydrate oxidation (g) and fat oxidation (g) measured via indirect calorimetry
Change in diet respiratory exchange ratio (RER) from baseline to 8 weeks | Measured at fasting and for 3.5h postprandially at baseline and 8 weeks
  RER measured via indirect calorimetry
Change in fasting and postprandial lipid peroxidation from baseline to 8 weeks | Measured at fasting and for 4 hours postprandially at baseline and 8 weeks
  Malondialdehyde (MDA) (uM) measured via Thiobarbituric acid reactive substances (TBARS) assay.
Change in fasting and postprandial total antioxidant capacity from baseline to 8 weeks | Measured at fasting and for 4 hours postprandially at baseline and 8 weeks
  Total antioxidant capacity (uM trolox equivalents) measured via Oxygen Radical Absorbance Capacity (ORAC) assay.
Changes in fasting and postprandial hunger and satiety from baseline to 8 weeks | Measured at fasting and for 4 hours postprandially at baseline and 8 weeks. Also, measured once per hour after the baseline and 8-week visits.
  Hunger, fullness, prospective consumption, and desire to eat measured via a Visual Analog Scale (VAS) (mm). The range of scores on the continuous VAS is 0-100 mm. Zero represents no hunger, fullness, prospective consumption, and desire to eat, while 100 represents the greatest feeling of these outcomes.

OTHER OUTCOMES:
Change in baseline perceived stress at 4 and 8 weeks | Baseline, 4 weeks, 8 weeks
  The perceived stress scale (PSS) measures stress over the last 4 weeks on a scale from 0-40. Low scores indicate low stress. A score of 13 is average. Scores of 20 or greater are considered to be high stress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Georgia- Department of Foods and Nutrition, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The plan is to share group averages through publication.

REFERENCES:
- [Derived] Guarneiri LL, Paton CM, Cooper JA. Pecan-Enriched Diets Alter Cholesterol Profiles and Triglycerides in Adults at Risk for Cardiovascular Disease in a Randomized, Controlled Trial. J Nutr. 2021 Oct 1;151(10):3091-3101. doi: 10.1093/jn/nxab248. PMID 34383903